CLINICAL TRIAL: NCT01223820
Title: Neuro-immunological Analysis of Idiopathic Rhinitis Patients and Controls Treated With Capsaicin.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, MD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nasal Capsaicin treatment
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Idiopathic Rhinitis Patients; Healthy Controls
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capsaicin (Experimental)
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin — 5x nasal application in one day, 1 hour between each application

SUMMARY:
The term idiopathic rhinitis (IR) is used in this study to describe a patient group with following characteristics: patients with complaints of nasal obstruction, sneezing and/or rhinorrhea for a period of over 1 year, which cannot be attributed to allergy, nasal or paranasal infection, anatomical disorders, pregnancy or lactation and/or systemic disorders. These patients are non-smokers and do not use medication affecting nasal function. They have no beneficial effect of intranasal steroid spray (INS) treatment.

The population incidence of IR is estimated to be as high as 10%. The pathophysiology of IR is largely unknown. Several hypotheses have been put forward. In general it is assumed that neurogenic mechanisms play an important role. Neuropeptides like CGRP, SP, NKA/B, NPY, NGF are released from afferent neurons in the nasal mucosa after activation by unspecific stimuli and can be responsible for the symptoms of IR.

For this group of IR-patients, there is until now only one treatment option: intranasal capsaicin application. Capsaicin, the pungent agent in hot pepper, is supposed to exert its' therapeutic effect via degeneration or desensitization effect on the afferent C-fibers.

The hypothesis is that nasal capsaicin treatment reduces neurogenic inflammation and reduces in that way nasal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent (> 12w) rhinological symptoms: nasal discharge, sneezing, congestion for an average of at least 1 h per day for at least 5 days during a period of 14 days, negative skin prick test or negative RAST, and without structural abnormalities explaining nasal obstruction will be proposed to participate in the trial.
2. Age > 18 and < 50 years
3. Written informed consent
4. Willingness to adhere to visit schedules
5. Adequate contraceptive precautions in female patients with childbearing potential
6. Unresponsiveness to nasal steroid spray (4 weeks of use)

Exclusion Criteria:

1. Age < 18 and > 50 years
2. Patients with AR, demonstrated by either positive skin prick test or RAST
3. Presence of IgE in nasal lavage fluid
4. Structural abnormalities: nasal polyps, severe septal deviation (septum reaching concha inferior or lateral nasal wall.
5. Systemic steroid treatment less than 4 weeks before the inclusion in the study.
6. Nasal steroid spray less than 4 weeks before the inclusion, oral leukotriene antagonists or long-acting antihistamines less than 2 weeks before the inclusion.
7. Inability of the patient to stop taking medication affecting nasal function.
8. Evidence of infectious rhinitis/rhinosinusitis.
9. Pregnancy or breastfeeding.
10. Any disorder of which might compromise the ability of a patient to give truly informed consent for participation in this study.
11. Enrollment in other investigational drug trial(s) or is receiving other investigational agent(s) for any other medical condition.
12. Contra-indications for local anaesthesia (Cocaïne 5%).
13. Smoking.
14. Systemic disease with lesions in ENT domain.
15. Malignancies or severe comorbidity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Neuro-immunological effect. | 6 months
  The primary aim of the study is to identify the neuro-immunological effects induced by capsaicin nasal spray in IR patients and healthy individuals.

SECONDARY OUTCOMES:
TR-PNIF-CDA | 7 months
  The secondary aim of this study is to correlate the neuro-immunological findings with the therapeutic response to capsaicin, the nasal congestion using the peak nasal inspiratory (PNIF), and nasal response to Cold Dry Air (CDA)-provocation.

CONTACTS AND LOCATIONS:
Overall Officials: Laura H Van Gerven, MD, Principal Investigator — UZ Leuven; Peter W Hellings, MD, PhD, Study Director — UZ Leuven
Locations (1):
- UZ Leuven, NKO-GH Kapucijnenvoer 33, Leuven, Vlaams-Brabant, Belgium